CLINICAL TRIAL: NCT01706146
Title: Rhythm Evaluation for AntiCoagulaTion With COntinuous Monitoring
Acronym: REACT COM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Medtronic (Industry)
Responsible Party: Principal Investigator, Alexandru B Chicos, Director, Cardiac Electrophysiology Laboratory Bluhm Cardiovascular Institute, Northwestern Memorial Hospital, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STU00064217; 1R34HL113404-01 (NIH); 7R34HL113404-03 (NIH)
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; reveal xt; oral anticoagulation; dabigatran; rivaroxaban; apixaban
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran; Rivaroxaban; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Non-Coumadin Oral Anticoagulant (Other): Administration of Non-coumadin Oral Anticoagulant for 30 days following episode of atrial fibrillation as detected by the Reveal XT device.
  Interventions: Drug: Non-coumadin Oral Anticoagulant

INTERVENTIONS:
Drug: Non-coumadin Oral Anticoagulant — Administration of Non-coumadin Oral Anticoagulant for 30 days following episode of atrial fibrillation as detected by the Reveal XT device.
  Other Names: Including but not limited to:; Dabigatran (Pradaxa); Rivaroxaban (Xarelto); Apixaban (Eliquis)

SUMMARY:
Atrial fibrillation (AF) is the most common sustained abnormal rhythm of the heart, affects an estimated 2.5 to 5 million individuals in the US, and can lead to stroke, heart failure, and premature death. For those with AF and other stroke risk factors, chronic anticoagulation is recommended to prevent intracardiac thrombus formation and stroke even if the AF is infrequent or short-lived. This standard of care is based partly on our inability to rapidly recognize and respond to AF recurrences which can often be brief and asymptomatic, but exposes the patient to the risk of anticoagulant-induced hemorrhage even during prolonged periods of sinus rhythm where the risk of stroke is presumably low.

Recent advances in device technology and drug therapy, however, have the potential to change the way the investigators manage AF. The use of a small leadless subcutaneous implantable cardiac monitor with remote data transmission capabilities (Reveal XT, Medtronic Inc.) provides the ability to remotely and continuously evaluate a patient for AF recurrences, even episodes that are brief and asymptomatic. In addition, release of unique oral thrombin inhibitor approved for use in non-valvular AF(Dabigatran [Pradaxa], Rivaroxaban [Xarelto]) allows for rapid onset anticoagulation within minutes to hours of a single oral dose. Together, these advances allow for continuous AF monitoring with targeted anticoagulation only around the time of an AF episode, thereby reducing the risk of drug-induced hemorrhage while still protecting against stroke.

The aim of this pilot study is to assess the feasibility of intermittent anticoagulation with a rapid-onset oral thrombin inhibitor guided by a continuous AF-sensing implantable cardiac monitor (Reveal XT) with remote data transmission capabilities.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria:

1. Age 18 and above.
2. Patients with non-valvular, non-continuous AF and either:

   (A) Infrequent AF episodes without a rhythm control strategy who have had no documented AF lasting > 1 hour for 3 consecutive months (the last 2 of which are on a previously implanted Reveal XT implantable cardiac monitor), or (B) Previous or current rhythm control strategy. Rhythm control strategies may include: i. Class I or Class III antiarrhythmic drugs ii. Pulmonary vein isolation iii. Post-MAZE/minimally invasive MAZE
3. Current Reveal XT implant prior to study enrollment.
4. Documented clinical history of symptomatic or asymptomatic paroxysmal, long-standing persistent or persistent AF prior to rhythm control initiation. The duration of AF must have been > 30 seconds as documented by an external monitor, present 12 lead ECG, or Reveal XT.
5. CHADS2 score of 1 or 2
6. Candidates for chronic anticoagulation with an FDA-approved non-Coumadin oral anticoagulant (dabigatran, rivaroxaban, apixaban), based on the discretion of the treating physician.
7. Demonstrated ability to tolerate dabigatran 150mg/BID (if CrCl >30ml/min), rivaroxaban 15mg QD (if CrCl 15-49 ml/min) and 20mg QD (if CrCl ≥50ml/min), or apixaban 5mg BID or 2.5 mg for subjects with ≥2 of the following: age ≥ 80 years, body weight ≤60kg, serum creatinine ≥1.5 mg/dl.
8. Able and willing to provide written informed consent and willing to follow instructions, attend all required study visits, and undergo all planned tests.
9. Subject must be willing and able to discontinue oral anticoagulation for the purposes of this study

Exclusion Criteria:

Patients should not have any of the following criteria:

1. Permanent AF
2. Any documented single AF episode lasting ≥ 1 hour per month over two consecutive months prior to study enrollment.

   Mechanical prosthetic valves or severe valve disease.
3. CHADS2 score of 0, or > 2
4. Subject deemed high risk for non-cardioembolic stroke (i.e. significant carotid artery disease) based on discretion of the investigator.
5. Individual is pregnant, nursing, or planning to become pregnant.
6. Known hypersensitivity to non-Coumadin oral anticoagulants.
7. Documented prior stroke or transient ischemic attack.
8. Reversible causes of AF (e.g., cardiac surgery, pulmonary embolism, untreated hyperthyroidism).
9. Conditions associated with an increased risk of bleeding:

   * Major surgery in the previous month
   * Planned surgery or intervention in the next 3 months.
   * History of intracranial, intraocular, spinal, retroperitoneal or atraumatic intra-articular bleeding
   * Gastrointestinal hemorrhage within the past year unless the cause has been permanently eliminated (e.g. by surgery)
   * Symptomatic or endoscopically documented gastroduodenal ulcer disease in the previous 30 days
   * Hemorrhagic disorder or bleeding diathesis
   * Need for anticoagulant treatment for disorders other than AF
   * Required use of non-aspirin antiplatelet agents (i.e., Plavix) at time of enrollment
   * Uncontrolled hypertension (SBP >180 mmHg and/or DBP >100 mmHg)
10. Recent malignancy or radiation therapy (≤6 months)
11. Anemia (hemoglobin <10g/dL) or thrombocytopenia (platelet count <100K/UL)
12. Patients who have received an investigational drug in the past 30 days or are participating in a drug study.
13. Intolerance or hypersensitivity to low dose aspirin therapy
14. Life expectancy less than the expected duration of the trial due to concomitant disease.
15. Any concomitant condition which, in the opinion of the investigator, would not allow safe participation in the study (e.g., drug addiction, alcohol abuse).
16. Inability to comply with daily data transmission requirements.
17. Known history of isolated atrial flutter/atrial tachycardia without atrial fibrillation.
18. More than 10 false positive atrial fibrillation events lasting > 30 minutes per month for two months prior to enrollment on a previously implantable cardiac monitor.
19. Severe renal impairment (CrCl < 15 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Chicos, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
- University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Derived] Passman R, Leong-Sit P, Andrei AC, Huskin A, Tomson TT, Bernstein R, Ellis E, Waks JW, Zimetbaum P. Targeted Anticoagulation for Atrial Fibrillation Guided by Continuous Rhythm Assessment With an Insertable Cardiac Monitor: The Rhythm Evaluation for Anticoagulation With Continuous Monitoring (REACT.COM) Pilot Study. J Cardiovasc Electrophysiol. 2016 Mar;27(3):264-70. doi: 10.1111/jce.12864. Epub 2015 Nov 23. PMID 26511221

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Coumadin Oral Anticoagulant
Started | 59
Completed | 53 (1 pt developed permanent AF; 1 pt needed dual antiplatelet therapy; 3 possible TIA; 1 withdraw)
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 3
Not completed — Developed AF and need for antiplatelets | 2

BASELINE CHARACTERISTICS:
Arm/Group | Non-Coumadin Oral Anticoagulant
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 38
Age, Continuous [Mean (Standard Deviation); unit: year] | 66.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 12
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Days on Anticoagulation
Description: Assess subject anticoagulant utilization and number of days on anticoagulation
Time Frame: up to 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Non-Coumadin Oral Anticoagulant
Number analyzed (Participants) | 59
days | 24.9 (51.9)

2. Secondary Outcome: Bleeding Incidence
Description: To assess the bleeding incidence with implantable monitor-guided intermittent anticoagulation.
Time Frame: up to 12 months
Measure: Number; unit: participants
Arm/Group | Non-Coumadin Oral Anticoagulant
Number analyzed (Participants) | 59
participants | 3

3. Other Pre Specified Outcome: Stroke Rate
Description: To assess the stroke rate with implantable monitor-guided intermittent anticoagulation.
Time Frame: 12 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Overall Survival
Description: To assess the overall survival rate with implantable monitor-guided intermittent anticoagulation.
Time Frame: 12 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Major Bleeding-free Survival Rate
Description: To assess the major bleeding-free survival rate with implantable monitor-guided intermittent anticoagulation.
Time Frame: 12 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Stroke-free Survival Rate
Description: To assess the stroke-free survival rate with implantable monitor-guided intermittent anticoagulation.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Non-Coumadin Oral Anticoagulant
Serious Adverse Events (participants affected / at risk) | 3/59
Other Adverse Events (participants affected / at risk) | 3/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Coumadin Oral Anticoagulant (N=59)
TIA (Nervous system disorders) | 3 (3) — There were 3 possible TIA events. Adjudication of the three potential TIA events by an independent review committee rated two as "possible TIA" and one as "definite TIA".
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Coumadin Oral Anticoagulant (N=59)
Minor bleeding (Vascular disorders) | 3 — There were two major bleeds following trauma, both occurring on aspirin therapy. Three minor bleeds occurred, two of which occurred on aspirin and one gastrointestinal bleed on NOAC.
Major Bleeding (Vascular disorders) | 2 (2) — There were two major bleeds following trauma, both occurring on aspirin therapy. Three minor bleeds occurred, two of which occurred on aspirin and one gastrointestinal bleed on NOAC
Development of Permanent Atrial Fibrillation (Cardiac disorders) | 1 (1) — One participant developed permanent AF.
Dual antiplatelet therapy (Blood and lymphatic system disorders) | 1 (1) — One participant required dual antiplatelet therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No